CLINICAL TRIAL: NCT02164929
Title: A Prospective, Randomized, Single-Blind Study to Evaluate the Efficacy of Transversus Abdominis Plane Versus Paravertebral Regional Blockade in Patients Undergoing Laparoscopic Colectomy
Brief Title: Comparison Study of Transversus Abdominal Plane, Paravertebral and Epidural Blocks in Laparoscopic Colectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00047810
Record Dates: First submitted 2014-06-11; First posted 2014-06-17 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-01

CONDITIONS: Laparoscopic Colorectal Resection
Keywords: TAP block; Paravertebral block; Epidural; Laparoscopic colectomy
MeSH Terms: interventions — Injections, Epidural; Acetaminophen; Dexamethasone; Propofol; Lidocaine; Epinephrine; Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Paravertebral block (Active Comparator): Bilateral PVB will be placed between T7-T10 interspaces preoperatively. Patients will be in a sitting position which allows easy identification of landmarks, and the patients are often more comfortable. Ultrasound will be used to identify the paravertebral space. At the appropriate dermatome under aseptic precautions, the needle (22-gauge, 8-10-cm short beveled spinal needle) will inserted 2.5-3 cm lateral to the most cephalad aspect of the spinous process and advanced perpendicular to the skin in all planes to contact the transverse process 3 of the vertebra below at a variable depth (2-4 cm). A 10 mL ropivacaine 0.25% will be injected at both T7 and T9 levels on each side (40 mL in total).
  Interventions: Procedure: Paravertebral block; Drug: Acetaminophen 1g IV; Drug: Dexamethasone 4mg; Drug: Midazolam up to 2mg; Drug: Propofol 1-2.5 mg/kg; Drug: Sevoflurane to keep a bispectral index of between 40-60; Drug: Local infiltration with 10 mL of plain ropivacaine 0.25%
- TAP block (Active Comparator): Bilateral posterior and subcostal TAP blocks guided by ultrasound will be performed in the preoperative holding area. A total of 80 mL ropivacaine 0.25% (4 injections, 20 mL per injection) will be injected evenly upon identification of the appropriate planes. In the event the placement of block is uncomfortable for the patients, it will be performed after induction of anesthesia. This approach is currently practiced in the OR. Extent and degree of anesthetic blockage will be measured using a 5-point sensation scale following the procedure at 4 areas on the anterior abdominal wall (above and below the umbilicus bilaterally).
  Interventions: Procedure: TAP block; Drug: Acetaminophen 1g IV; Drug: Dexamethasone 4mg; Drug: Midazolam up to 2mg; Drug: Propofol 1-2.5 mg/kg; Drug: Sevoflurane to keep a bispectral index of between 40-60; Drug: Local infiltration with 10 mL of plain ropivacaine 0.25%
- Epidural (Active Comparator): An epidural catheter will be inserted between T8-10 in the preoperative holding area, and a test dose of 1.5% lidocaine with 1:200,000 epinephrine will be given. Extent and degree of anesthetic blockage will be measured using a 5-point sensation following the procedure and postoperatively at 4 areas on the anterior abdominal wall (above and below the umbilicus bilaterally).
  A bolus does of epidural hydromorphone (400-800 mcg) will be given preoperatively. An infusion of bupivacaine 0.25% at 4-6 ml/hour will be commenced before incision, and if tolerated, continued throughout surgery. Adjustments that may be required secondary to specific patient hemodynamic status will be left to the discretion of the individual anesthesiologist and guided by the specific patient requirements.
  Interventions: Procedure: Epidural; Drug: Acetaminophen 1g IV; Drug: Dexamethasone 4mg; Drug: Midazolam up to 2mg; Drug: Propofol 1-2.5 mg/kg; Drug: Sevoflurane to keep a bispectral index of between 40-60; Drug: Local infiltration with 10 mL of plain ropivacaine 0.25%; Drug: Lidocaine; Drug: Epinephrine; Drug: Hydromorphone
- No block (PCA alone) (Active Comparator): Premedication with midazolam up to 2 mg. General anesthesia is induced with propofol 1-2.5 mg/kg. Dexamethasone 4 mg IV will be administered after induction of anesthesia. Anesthesia will be maintained with sevoflurane to keep a bispectral index of between 40-60. Neuromuscular blocking drug and reversal agent of choice may be used. Local infiltration with 10 mL of plain ropivacaine 0.25% will be administered at the surgical incision site at the end of surgery. Acetaminophen 1g IV will be administered following induction of anesthesia will be administered at the end of the procedure
  Interventions: Drug: Acetaminophen 1g IV; Drug: Dexamethasone 4mg; Drug: Midazolam up to 2mg; Drug: Propofol 1-2.5 mg/kg; Drug: Sevoflurane to keep a bispectral index of between 40-60; Drug: Local infiltration with 10 mL of plain ropivacaine 0.25%

INTERVENTIONS:
Procedure: TAP block
  Other Names: Transversus abdominus plane block
  Arms: TAP block
Procedure: Epidural
  Other Names: Thoracic Epidural Anesthesia (TEA)
  Arms: Epidural
Procedure: Paravertebral block
  Other Names: PVB
  Arms: Paravertebral block
Drug: Acetaminophen 1g IV
Drug: Dexamethasone 4mg
Drug: Midazolam up to 2mg
Drug: Propofol 1-2.5 mg/kg
Drug: Sevoflurane to keep a bispectral index of between 40-60
Drug: Local infiltration with 10 mL of plain ropivacaine 0.25%
Drug: Lidocaine — 1.5% lidocaine
  Arms: Epidural
Drug: Epinephrine — 1:200,000 epinephrine
  Arms: Epidural
Drug: Hydromorphone — 400-800 mcg Hydromorphone will be given preoperatively
  Arms: Epidural

SUMMARY:
The purpose of this study is to assess the effectiveness of transversus abdominal plane (TAP) block, thoracic epidural or paravertebral block (PVB) for controlling postoperative pain when compared with opioid you self-administer in your vein using a PCA device. The primary outcome will be postoperative opioid consumption within 24 hours after surgery. A total of 120 subjects will be randomized in a 1:1:1:1 ratio to receive a TAP block, PVB, TEA or no block (PCA alone).Patients in all groups will be cared for using an established enhanced recovery after surgery (ERAS) pathway incorporating a multimodal analgesic regimen using IV acetaminophen and postoperative PCA fentanyl.

ELIGIBILITY:
Inclusion Criteria

* Male or female, ≥ 18 years of age
* Patients scheduled to undergo laparoscopic colectomy without stoma under general anesthesia
* American Society of Anesthesiology (ASA) Physical Class 1-3.

Exclusion Criteria:

* Open colectomy
* Perineal resection
* Stoma formation
* Patients with a contraindication to TEA or regional anesthesia.
* Pregnancy, nursing, or planning to become pregnant during the study or within one month.
* Long-acting opioid medication within 3 days.
* Any opioid medication within 24 hours.
* Body weight less than 50 kilograms (~110 pounds)
* Uncontrolled anxiety, schizophrenia, or other psychiatric disorder
* Current or historical evidence of any clinically significant disease or condition that, in the opinion of the Investigator, may increase the risk of surgery or complicate the subject's postoperative course.
* Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.
* Suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
* Significant medical conditions or laboratory results that, in the opinion of the Investigator, indicate an increased vulnerability to study drugs and procedures, and expose the subject to an unreasonable risk as a result of participating in this clinical trial, such as: debilitating diseases, acute illnesses, hypotension, partial or complete conduction block, impaired cardiac function, untreated hypertension, advanced arteriosclerotic heart disease, cerebral vascular insufficiency, pre-existing abnormal neurological or neuromuscular disease (e.g., epilepsy, myasthenia gravis), advanced liver disease, severe renal impairment, advanced diabetes, comorbid conditions associated with an immunocompromised status, such as blood dyscrasias, HIV/AIDS, or recent chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 17 patients that consented, one patient withdrew before randomization
Groups:
- Paravertebral Block: Bilateral PVB will be placed between T7-T10 interspaces preoperatively. Patients will be in a sitting position which allows easy identification of landmarks, and the patients are often more comfortable. Ultrasound will be used to identify the paravertebral space. At the appropriate dermatome under aseptic precautions, the needle (22-gauge, 8-10-cm short beveled spinal needle) will inserted 2.5-3 cm lateral to the most cephalad aspect of the spinous process and advanced perpendicular to the skin in all planes to contact the transverse process 3 of the vertebra below at a variable depth (2-4 cm). A 10 mL ropivacaine 0.25% will be injected at both T7 and T9 levels on each side (40 mL in total).
  Paravertebral block
  Acetaminophen 1g IV
  Dexamethasone 4mg
  Midazolam up to 2mg
  Propofol 1-2.5 mg/kg
  Sevoflurane to keep a bispectral index of between 40-60
  Local infiltration with 10 mL of plain ropivacaine 0.25%
- TAP Block: Bilateral posterior and subcostal TAP blocks guided by ultrasound will be performed in the preoperative holding area. A total of 80 mL ropivacaine 0.25% (4 injections, 20 mL per injection) will be injected evenly upon identification of the appropriate planes. In the event the placement of block is uncomfortable for the patients, it will be performed after induction of anesthesia. This approach is currently practiced in the OR. Extent and degree of anesthetic blockage will be measured using a 5-point sensation scale following the procedure at 4 areas on the anterior abdominal wall (above and below the umbilicus bilaterally).
  TAP block
  Acetaminophen 1g IV
  Dexamethasone 4mg
  Midazolam up to 2mg
  Propofol 1-2.5 mg/kg
  Sevoflurane to keep a bispectral index of between 40-60
  Local infiltration with 10 mL of plain ropivacaine 0.25%
- Epidural: An epidural catheter will be inserted between T8-10 in the preoperative holding area, and a test dose of 1.5% lidocaine with 1:200,000 epinephrine will be given. Extent and degree of anesthetic blockage will be measured using a 5-point sensation following the procedure and postoperatively at 4 areas on the anterior abdominal wall (above and below the umbilicus bilaterally).
  A bolus does of epidural hydromorphone (400-800 mcg) will be given preoperatively. An infusion of bupivacaine 0.25% at 4-6 ml/hour will be commenced before incision, and if tolerated, continued throughout surgery. Adjustments that may be required secondary to specific patient hemodynamic status will be left to the discretion of the individual anesthesiologist and guided by the specific patient requirements.
  Epidural
  Acetaminophen 1g IV
  Dexamethasone 4mg
  Midazolam up to 2mg
  Propofol 1-2.5 mg/kg
  Sevoflurane to keep a bispectral index of between 40-60
  Local infiltration with 10 mL of plain ropi
- No Block (PCA Alone): Premedication with midazolam up to 2 mg. General anesthesia is induced with propofol 1-2.5 mg/kg. Dexamethasone 4 mg IV will be administered after induction of anesthesia. Anesthesia will be maintained with sevoflurane to keep a bispectral index of between 40-60. Neuromuscular blocking drug and reversal agent of choice may be used. Local infiltration with 10 mL of plain ropivacaine 0.25% will be administered at the surgical incision site at the end of surgery. Acetaminophen 1g IV will be administered following induction of anesthesia will be administered at the end of the procedure
  Acetaminophen 1g IV
  Dexamethasone 4mg
  Midazolam up to 2mg
  Propofol 1-2.5 mg/kg
  Sevoflurane to keep a bispectral index of between 40-60
  Local infiltration with 10 mL of plain ropivacaine 0.25%
Period: Overall Study
Arm/Group | Paravertebral Block | TAP Block | Epidural | No Block (PCA Alone)
Started | 4 | 3 | 5 | 4
Completed | 3 | 3 | 4 | 2
Not Completed | 1 | 0 | 1 | 2
Not completed — Converted to open procedure | 1 | 0 | 0 | 2
Not completed — Failed regional block | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants that completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Paravertebral Block | TAP Block | Epidural | No Block (PCA Alone) | Total
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (8.5) | 51 (15) | 57.75 (6.6) | 52 (21.9) | 54.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 2 | 7
  Male | 2 | 2 | 2 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Opioid Consumption
Description: If opioid other than fentanyl is used, the dose will be converted to morphine equivalent.
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Paravertebral Block | TAP Block | Epidural | No Block (PCA Alone)
Number analyzed (Participants) | 3 | 3 | 4 | 2
mcg | 734 (422) | 666 (474) | 125 (50) | 1017.5 (484)

2. Secondary Outcome: Pain Scores
Description: Pain scores at rest and with activity using a verbal rating scales (VRS) of 0-10, where "0" represents no pain and "10" represents worst pain ever, at 30, 60, 90, 120 min and every 6 hours for 24 hours and every 12 hours for 48 hours and once a day thereafter until discharge. Data were collected at the indicated time points and an average pain score was calculated.
Time Frame: Participants will be followed for the duration of hospital stay, an estimated 1 week
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paravertebral Block | TAP Block | Epidural | No Block (PCA Alone)
Number analyzed (Participants) | 3 | 3 | 4 | 2
Units on a scale | 4.66 (1.15) | 2.66 (1.52) | 1.75 (1.25) | 6 (2.82)

3. Secondary Outcome: Quality of Recovery
Description: Quality of Recovery Score (QoR-15) is measured on a scale of 0-150 (0=poor, 150 = excellent). Scores were collected daily for 72 hours and then averaged.
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paravertebral Block | TAP Block | Epidural | No Block (PCA Alone)
Number analyzed (Participants) | 3 | 3 | 4 | 2
Units on a scale | 89.5 (10.6) | 117 (23.3) | 115.5 (0.7) | 99 (17.6)

4. Secondary Outcome: Complications as Measured by a Modified Postoperative Morbidity Survey (MPMS)
Description: Complications using a Modified Postoperative Morbidity Survey (MPMS)
Time Frame: Participants will be followed for the duration of hospital stay, an estimated 1 week
Population: Data not collected
Arm/Group | Paravertebral Block | TAP Block | Epidural | No Block (PCA Alone)
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Time to First Bowel Movement
Time Frame: Participants will be followed for the duration of hospital stay, an estimated 1 week
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Paravertebral Block | TAP Block | Epidural | No Block (PCA Alone)
Number analyzed (Participants) | 3 | 3 | 4 | 2
days | 1 (1.4) | 2 (0.7) | 1 (0.8) | 2 (0)

6. Secondary Outcome: Opioid Related Side Effects
Description: Occurrence and duration of opioid related adverse events including postoperative nausea and vomiting (PONV); pruritus, urinary retention, confusion, sedation and respiratory depression at the above time points.
Time Frame: Participants will be followed for the duration of hospital stay, an estimated 1 week
Measure: Number; unit: side effects
Arm/Group | Paravertebral Block | TAP Block | Epidural | No Block (PCA Alone)
Number analyzed (Participants) | 3 | 3 | 4 | 2
side effects | 0 | 0 | 0 | 0

7. Secondary Outcome: Time to First Ingestion of Solid Food
Time Frame: Participants will be followed for the duration of hospital stay, an estimated 1 week
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Paravertebral Block | TAP Block | Epidural | No Block (PCA Alone)
Number analyzed (Participants) | 3 | 3 | 4 | 2
Days | 1 (0) | 2 (0.7) | 0.75 (0.5) | 1.5 (0.7)

8. Secondary Outcome: Number of Epidural-related Side Effects
Time Frame: Participants will be followed for the duration of hospital stay, an estimated 1 week
Measure: Number; unit: Number of side effects
Arm/Group | Paravertebral Block | TAP Block | Epidural | No Block (PCA Alone)
Number analyzed (Participants) | 3 | 3 | 4 | 2
Number of side effects | 0 | 0 | 0 | 0

9. Secondary Outcome: Length of Stay
Time Frame: Participants will be followed for the duration of hospital stay, an estimated 1 week
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Paravertebral Block | TAP Block | Epidural | No Block (PCA Alone)
Number analyzed (Participants) | 3 | 3 | 4 | 2
Days | 2.66 (0.57) | 4.33 (3.21) | 4 (1.41) | 3.5 (0.7)

ADVERSE EVENTS:
Arm/Group | Paravertebral Block | TAP Block | Epidural | No Block (PCA Alone)
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes